CLINICAL TRIAL: NCT05108792
Title: Continuous Deep Sedation Until Death Following a Decision to Limit or Stop Treatment in Intensive Care and in Continuous Surveillance Units
Brief Title: Continuous Deep Sedation Until Death
Acronym: SPCMD-REA
Status: Completed | Type: Observational
Sponsor: Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Sponsor
Other Study IDs: SPCMD-REA / NR 2020-01
Record Dates: First submitted 2021-10-14; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Terminal Care
Keywords: Limit or Stop Treatment in Intensive Care; Continuous deep sedation (CDS); Continuous deep sedation until death (CDSUD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients deceased following a decision to limit or stop therapeutics: a
  Interventions: Other: NO INTERVENTION

INTERVENTIONS:
Other: NO INTERVENTION — observational study, no intervention performed

SUMMARY:
This research is a descriptive observational study conducted in multicenter (intensive care and continuing care units) in France. All data collected is part of the patient record. The main objective is to describe the end-of-life sedative practices following a decision to limit or stop therapy in intensive care unit and continuing care unit.

DETAILED DESCRIPTION:
All participating sites will include last 10 consecutive major patients deceased following a decision to limit or stop therapeutics. The study include only data from patients died before January 1, 2020. In the case report form the following information will be entered:

* the characteristics of the unit of intensive care or continuing care unit.
* Patient Characteristics
* Characteristics of sedative practices

ELIGIBILITY:
Inclusion Criteria:

* Adult patients at the time of death (>18years)
* Died in intensive care or in continuing care unit
* Patient died before January 1st, 2020.
* Patients deceased following a decision to limit or stop therapeutics

Exclusion Criteria:

* Patients who died of brain death or unexpected cardiac arrest at death of unsuccessful cardiopulmonary resuscitation
* Patient who expressed during his lifetime his opposition to the use of his data for scientific research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients at the time of death (>18years) Died in intensive care or in continuing care unit following a decision to limit or stop therapeutics
Sampling Method: Probability Sample
Enrollment: 585 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Description of end-of-life sedative practices | after patient death (before january 1st 2020)
  Information concerning end-of-life sedative practices are recorder in the CRF (treatments used, patient's and unit characteristics...)

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu LE DORZE, MD, Study Chair — GH Lariboisière-St Louis
Locations (64):
- France (64):
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CH Arras, Arras
  - CHR Metz Thionville, Ars-Laquenexy
  - CH Henri Mondor d'Aurillac, Aurillac
  - CHU Jean Minjoz, Besançon
  - Centre Hospitalier de Chateau Thierry, Château-Thierry
  - Hôpital d'Instruction des Armées Percy, Clamart
  - CHU Clermont-Ferrand - Site de Gabriel Montpied - Neuroréanimation, Clermont-Ferrand
  - CHU Clermont-Ferrand - Site de Gabriel Montpied - Réa médico chir, Clermont-Ferrand
  - Hôpital Beaujon - Réa hépato digestive, Clichy
  - Hôpital Beaujon - Réa neuro chir, Clichy
  - CH de DAX, Dax
  - CHU de Grenoble - Hôpital A Michallon, Grenoble
  - Hôpital privé de Marne la Vallée, Jossigny
  - Groupe Hospitalier LITTORAL ATLANTIQUE, La Rochelle
  - Centre Hospitalier de Laon - Réanimation Polyvalente, Laon
  - CH de Versailles - André Mignot, Le Chesnay
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHRU de Lille - Réa Neurochirurgicale, Lille
  - CHRU de Lille - service de déchocage et de soins intensifs - Urgence, Lille
  - CHRU de Lille- Hôpital Huriez, Lille
  - CHU la Timone 2 - Pôle GEST - RUSH, Marseille
  - Hôpital Nord Aphm, Marseille
  - CH Mont de Marsan, Mont-de-Marsan
  - Centre Hospitalier de Montélimar, Montélimar
  - CHU de Montpellier - Hopital Gui de Chauliac - Réa médicale, Montpellier
  - CHU de Montpellier - Hopital Gui de Chauliac, Montpellier
  - CHU MONTPELLIER - Hôpital Arnaud de Villeneuve, Montpellier
  - CHU Montpellier - Hôpital Lapeyronie, Montpellier
  - Groupe hospitalier de la région de Mulhouse et Sud-Alsace _ GHRMSA Mulhouse, Mulhouse
  - CHRU de NANCY, Nancy
  - CHU Nantes, Hôtel-Dieu, Nantes
  - Hôpital Pasteur 2 - CHU de Nice, Nice
  - Hôpital Privé Gériatrique Les Sources- Nice, Nice
  - CHU de Nimes, Nîmes
  - Centre Hospitalier territorial de Nouméa en Nouvelle Calédonie, Nouméa
  - Centre Hospitalier d'Orléans, Orléans
  - Centre Hospitalier Sainte-Anne, Paris
  - CHU Bichat Claude Bernard, Paris
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - Hôpital Lariboisière, Paris
  - Hôpital Pitié-Salpêtrière - Réa neuro chir, Paris
  - Hôpital Pitié-Salpêtrière - Réanimation Polyvalente, Paris
  - Hôpital Pitié-Salpêtrière Paris - SSPI, Paris
  - hôpital Saint Antoine - Paris, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Reims, Reims
  - CHU de Rennes - Réanimation chirurgicale, Rennes
  - CHU de Rennes - Réanimation CTCV, Rennes
  - Hôpitaux Drôme Nord - Site de Romans, Romans
  - CHU de Rouen, Rouen
  - CHU Rouen - Réanimation cardiaque chirurgicale, Rouen
  - Centre Hospitalier Privé Saint-Grégoire, Saint-Grégoire
  - CHRU Strasbourg, Strasbourg
  - Hôpital d'Instruction des Armées Sainte Anne, Toulon
  - CHU de Toulouse - Hôpital Pierre-Paul, Toulouse
  - CHU de Toulouse-Rangueil, Toulouse
  - CHU Rangueil - Toulouse - Réanimation de Néphrologie et Transplantation, Toulouse
  - Clinique Pasteur, Toulouse
  - CHRU Tours, Site Trousseau - Réa chir, Tours
  - CHRU Tours, Site Trousseau - URTC-B, Tours
  - Centre Hospitalier Bretagne Atlantique de Vannes, Vannes
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided